CLINICAL TRIAL: NCT01264731
Title: Combination Therapy of Topical Imiquimod Plus Multipeptide Vaccination for Cutaneous Metastases of Melanoma
Acronym: MEL53
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Craig L Slingluff, Jr, Professor of Surgery, Principal Investigator, University of Virginia Health System, Department of Surgery, Human Immune Therapy Center, University of Virginia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15168
Record Dates: First submitted 2010-12-20; First posted 2010-12-22 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Melanoma
Keywords: melanoma; peptide vaccine; aldara; imiquimod; immunotherapy
MeSH Terms: conditions — Melanoma | interventions — Imiquimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- peptide vaccine plus imiquimod (Active Comparator): Peptide Vaccine: Days 1, 8, 15, 36, 57, 78 Imiquimod: Applied daily on days 1-85.
  Interventions: Biological: MELITAC 12.1; Drug: Imiquimod
- Imiquimod (Active Comparator): Imiquimod: Applied daily on days 1-85.
  Interventions: Drug: Imiquimod

INTERVENTIONS:
Biological: MELITAC 12.1 — Vaccine regimen: The vaccines will be administered in two treatment cycles. During cycle one, three vaccines will be administered over a 3-week period on days 1, 8, and 15. During cycle two, three vaccines will be administered over a 9-week period on days 36, 57, 78. Participants in cohort 1 will receive MELITAC 12.1 (100 mcg each of the12-MP and 200 mcg of Peptide-tet) administered subcutaneously (1 ml) and intradermally (1 ml) in Montanide ISA-51 VG adjuvant at a single vaccination site.
  Arms: peptide vaccine plus imiquimod
Drug: Imiquimod — Topical Imiquimod regimen: Beginning on day 1, patients in cohorts 1 and 2 will have one or more cutaneous melanoma metastases treated topically with 5% imiquimod cream, with a dose of 1 to 3 packets of imiquimod daily, (depending on the extent of cutaneous metastases). Each packet contains 250 mg of cream and may be used for a surface area of up to 20 cm2. The number of lesions that are treated will be dependent on the availability and size of the lesions. In addition, if available, at least two lesions will be followed without treatment with the plan that they will be excised at week 3 (day 22) and week 6 (day 43), respectively, as controls. Imiquimod will be applied daily for seven days each week for 12 weeks. One course of treatment will be three weeks in duration, with evaluation by a clinician after every treatment course.
  Other Names: Aldara

SUMMARY:
The purpose of the study is to determine 1) the safety of administration of topical 5% imiquimod cream with or without administration of a peptide-based vaccine in patients with cutaneous metastases of melanoma and 2) evaluate whether topical imiquimod at sites of melanoma metastasis, with or without vaccine, increases a) endothelial expression of E-selectin and b) T cell infiltration.

DETAILED DESCRIPTION:
Primary goals:

Safety:

1) To determine the safety of administration of topical 5% imiquimod cream with or without administration of a peptide-based vaccine in patients with cutaneous metastases of melanoma.

Biologic effect:

1) To evaluate whether topical imiquimod at sites of melanoma metastasis, with or without vaccine, increases a) endothelial expression of E-selectin and b) T cell infiltration.

Secondary goals:

1. To assess whether T cells infiltrating melanoma metastases after imiquimod, with and without vaccination, are reactive to peptides in the vaccine.
2. To evaluate whether topical imiquimod decreases the proportion of FoxP3+ CD25hi CD4+ cells (putative regulatory T cells, Tregs) among tumor infiltrating T cells.
3. To estimate the effects of vaccine on CXCR3, CLA, and activation marker expression by circulating and tumor-infiltrating antigen-experienced CD4 and CD8 T cells.
4. To obtain preliminary data on the clinical response of cutaneous metastases of melanoma to the proposed combination regimen.
5. To determine the expression of TLR7 by immune cells and/or melanoma cells in the metastatic melanoma microenvironment.
6. To obtain preliminary data on associations between metastatic melanoma T cell infiltration patterns (immunotypes) and molecular and clinical responses to imiquimod.

Design:

The present proposal is for a clinical trial and associated correlative studies that bring together several observations and unmet scientific and clinical needs that have promise for a new effective immunotherapy for melanoma metastases. This is an open-label two-cohort, nonrandomized, pilot study of a combination of topical imiquimod plus systemic vaccination with MELITAC 12.1 vaccine, an emulsion of a mixture of 12 class I MHC-restricted melanoma peptides (12-MP) and a class II MHC-restricted tetanus toxoid helper peptide (tet). Cohort 1 will receive the combination of imiquimod + vaccine; Cohort 2 will receive imiquimod only. Patients will be eligible for cohort 1 if they are eligible for the vaccine based on HLA type and clinical factors. Cohort 2 is for patients who are not eligible for the vaccine.

Primary Endpoints:

Safety:

1) Toxicity profile of topical imiquimod at sites of melanoma, with or without MELITAC 12.1 vaccine.

Biologic effect:

1) Change in levels of intratumoral E-selectin and infiltrating TCD4 and TCD8 lymphocytes:

1. pretreatment vs after vaccine + imiquimod;
2. with vaccine vs. without vaccine (cohorts 1 vs 2);
3. lesions with imiquimod vs. without imiquimod.

Secondary Endpoints:

The following will be evaluated by comparing pretreatment to after vaccine + imiquimod, and comparing findings from patients with and without vaccine (cohorts 1 and 2), as well as lesions with and without imiquimod.

1. Change in the number of vaccine-reactive T cells in the melanoma metastases, as determined by ELIspot and tetramer analyses.
2. Change in the percentage of FoxP3+ CD25hi CD4+ (putative regulatory T cells, Tregs) among tumor infiltrating T cells as determined by immunohistochemistry and flow cytometry.
3. Expression of CXCR3, CLA, and activation markers (CD69, CD137, HLA-DR, CD27 and CD28) on vaccine-reactive cells in the blood and within the melanoma metastases by immunohistochemistry and flow cytometric analyses.
4. TLR7 expression by cells in the metastatic melanoma microenvironment.
5. Changes in T cell infiltration patterns of metastases (immunotype)

   The following will be evaluated post-treatment
6. Clinical regression of individual imiquimod-treated and untreated metastases

ELIGIBILITY:
Inclusion Criteria:

1. Participants with stage IIIB, IIIC or IV melanoma with cutaneous metastases.
2. Patients must have adequate cutaneous metastases of melanoma readily accessible for biopsy to provide a minimum of 0.3 cm3 of tissue per biopsy (approximately 0.85 cm by 0.85 cm x 0.85 cm or five 2mm core biopsies) at each of three time points. Several scenarios may fulfill the tumor burden requirement. For example, a patient may have one large lesion from which core biopsies can be taken for the first and second biopsy time points and then the entire lesion excised for the final tissue sample. Other combinations are acceptable.
3. The intent is to limit this study to patients with cutaneous melanoma metastasis rather than subcutaneous or lymph node metastasis because imiquimod may not penetrate to those deeper metastases.
4. Patients may have had multiple primary melanomas.
5. Patients may have had or may have a metastasis from a cutaneous primary site, mucosal primary site, ocular primary site, or unknown primary site.
6. Patients who have had brain metastases may be eligible if they meet the following criteria

   * Patients with less than or equal to 5 metastases may be eligible as long as the following 3 criteria are true:
   * The brain metastases have been completely removed by surgery or have been treated completely by stereotactic radiotherapy. Stereotactic radiotherapy, such as gamma knife, can be used up to 1 week prior to study entry.
   * There has been no evident growth of any brain metastasis since treatment.
   * No metastasis greater than 2 cm at the time of protocol entry
   * Patients with greater than 5 metastases may be eligible if the above 3 criteria are met and if at least one year has elapsed since the last treatment.
7. All participants must have ECOG performance status of 0 or 1 and ability and willingness to give informed consent
8. Patients must have at least one intact axillary and/or inguinal lymph node basin. A patient with a prior lymph node biopsy may be a candidate if lymphoscintigraphy demonstrates intact drainage to a node in that basin. A lymphoscintigram may be performed during screening to ensure that there is drainage to a regional node from a planned vaccine site. If the lymphoscintigram is performed and a sentinel lymph node is not located, the patient will be ineligible for this study if no other vaccine sites are available.
9. Laboratory parameters as follows: The following laboratory parameters will be required for all participants. If a lab value appears to be an error or a result of a transient or treatable condition, the investigator will use his/her clinical judgment to decide if the test may be repeated. The requirements for inclusion are as follows:

   * HLA-A1, -A2, -A3, or -A11+
   * ANC > 1000/mm3
   * Platelets > 100,000/mm3
   * Hgb ≥ 9 g/dL
   * HGBA1C < 7%
   * AST and ALT ≤ 2.5 x upper limits of normal (ULN)
   * Bilirubin ≤ 2.5 x ULN
   * Alkaline phosphatase ≤ 2.5 x ULN
   * Creatinine ≤ 1.5 x ULN
   * HIV negative (within 6 months of study entry)
   * Hepatitis C negative (within 6 months of study entry)
   * LDH up to 2 x ULN
10. Patients must be 18 years or older at study entry

Exclusion Criteria:

1. Patients who have had brain metastases unless they meet the criteria outlined above
2. Patients who are currently receiving systemic cytotoxic chemotherapy, radiation, or other experimental therapy, or who have received this therapy within the preceding 4 weeks. Gamma knife or stereotactic radiosurgery may be administered within the prior 4 weeks, but must not be administered less than one week prior to study enrollment. Patients who are currently receiving nitrosoureas or who have received this therapy within the preceding 6 weeks.
3. Patients will not be eligible if there is clinically detectable melanoma deemed likely by the investigator to require intervention during the first 12 weeks of the study that would require premature discontinuation. Examples for such circumstances may include untreated bone metastases at risk for fracture, and rapidly progressive low volume disease.
4. Patients with known or suspected allergies to any component of the vaccine.
5. Patients receiving the following medications at study entry or within the preceding 4 weeks are excluded:

   * Agents with putative immunomodulating activity (with the exception of non-steroidal anti-inflammatory agents and topical steroids
   * Allergy desensitization injections.
   * Systemic corticosteroids, administered parenterally or orally. Inhaled steroids (e.g. Advair®, Flovent®, Azmacort®) are not permitted. Topical corticosteroids are acceptable, including steroids with very low solubility administered nasally for local effects only (e.g. Nasonex®).
   * Any pharmacologic growth factors (e.g. GM-CSF, G-CSF, erythropoietin).
   * Interferon therapy.
   * Interleukin-2 or other interleukins.
   * Topical 5% Imiquimod cream: Patients must not have had imiquimod therapy to any body site within 4 weeks of study entry and must not have had any prior imiquimod therapy to the lesions to be treated, watched or biopsied on this present study. If imiquimod has been used in the past and either led to complete regression of the treated lesions, or those lesions have been removed surgically, then the patient may be eligible.
6. Prior melanoma vaccinations may be an exclusion criterion in som circumstances:

   * Patients who have recurred or progressed either after or during administration of a melanoma vaccine may be eligible to enroll 12 weeks following their last vaccination.
   * Patients may have been vaccinated previously with peptide vaccines (including MELITAC 12.1 and similar vaccines) or with non-peptide vaccines.
7. Pregnancy or the possibility of becoming pregnant during vaccine administration. Female patients of child-bearing potential must have a negative pregnancy test (urinary or serum beta-HCG) prior to administration of the first vaccine dose. Males and females must agree, in the consent form, to use effective birth control methods during the course of vaccination. Women must also not be breast feeding. This is consistent with existing standards of practice for vaccine and chemotherapy protocols.
8. Patients in whom there is a medical contraindication or potential problem in complying with the requirements of the protocol, in the opinion of the investigator.
9. Patients classified according to the New York Heart Association classification as having Class III or IV heart disease (Appendix 4).
10. Patients with a body weight < 110 lbs because of the amount and frequency with which blood will be drawn
11. Participants must not have had prior autoimmune disorders requiring cytotoxic or immunosuppressive therapy, or autoimmune disorders with visceral involvement. Participants with an active autoimmune disorder requiring these therapies are also excluded. The following will not be exclusionary:

    * The presence of laboratory evidence of autoimmune disease (e.g. positive ANA titer) without associated symptoms
    * Clinical evidence of vitiligo
    * Other forms of depigmenting illness
    * Mild arthritis requiring NSAID medications or no medical therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Safety: To determine the safety of administration of topical 5% imiquimod cream with or without administration of a peptide-based vaccine in patients with cutaneous metastases of melanoma. | 6 months

SECONDARY OUTCOMES:
Biologic: To evaluate whether topical imiquimod at sites of melanoma metastasis, with or without vaccine, increases a) endothelial expression of E-selectin and b) T cell infiltration. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Craig L Slingluff, M.D., Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

REFERENCES:
- [Derived] Tran CA, Lynch KT, Meneveau MO, Katyal P, Olson WC, Slingluff CL Jr. Intratumoral IFN-gamma or topical TLR7 agonist promotes infiltration of melanoma metastases by T lymphocytes expanded in the blood after cancer vaccine. J Immunother Cancer. 2023 Feb;11(2):e005952. doi: 10.1136/jitc-2022-005952. PMID 36746511